CLINICAL TRIAL: NCT00939081
Title: Community Based Obesity Prevention Among Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2794
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Obesity; Women's health; Minority health; Obesity prevention
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10,000 step/day recommendation (Active Comparator): Participants will receive a standard 10,000 step/day recommendation and 3 education sessions: at baseline, at 3 months and at 6 months.
  Interventions: Behavioral: 10,000 step/day recommendation
- Adaptive recommendation (Experimental): The adaptive recommendation will update the participant's recommended step count attainment from 7,000 to 8,000, then 10,000 steps/day. The SMS-based self-monitoring system will collect three data points each day from participants in this group: 1) total number of steps/d recorded by the pedometer during the previous day (steps/d); 2) performance on 2nd weight loss goal; and 3) performance on 3rd weight loss goal.
  Interventions: Behavioral: Adaptive step recommendation

INTERVENTIONS:
Behavioral: Adaptive step recommendation — Participants in this group receive 3 education sessions: at baseline, at 3 months and at 6 months. The adaptive recommendation will update the participant's recommended step count attainment from 7,000 to 8,000, then 10,000 steps/day. The SMS-based self-monitoring system will collect three data points each day from participants in this group: 1) total number of steps/d recorded by the pedometer during the previous day (steps/d); 2) performance on 2nd weight loss goal; and 3) performance on 3rd weight loss goal.
  Arms: Adaptive recommendation
Behavioral: 10,000 step/day recommendation — Participants will receive a standard 10,000 step/day recommendation and 3 education sessions: at baseline, at 3 months and at 6 months.
  Arms: 10,000 step/day recommendation

SUMMARY:
The purpose of this study is to examine whether pedometer step count recommendations (10,000 steps/day versus an adaptive recommendation) are differentially associated with the primary outcome of adherence to the pedometer-based physical activity regimen and the secondary outcomes of change in physical activity and body mass index (BMI).

DETAILED DESCRIPTION:
Long-term promotion of physical activity is necessary to achieve obesity prevention. This represents a particular challenge for our intervention design, as few studies have demonstrated positive long-term physical activity promotion outcomes among Black women. We have demonstrated the utility of pedometers among low income, ethnically diverse populations. The efficacy of pedometer utilization for the prevention of weight gain, however, hinges on long-term utilization of the devices. We hypothesize that recommendation for the step count attainment may affect individual's long-term utilization of pedometers, as well as physical activity levels and BMI.

This study is a 24-week experimental trial to examine whether intervention recommendations promote long-term adherence to a pedometer-based physical activity regimen. A two-group, block design will be used in the proposed study. Eligible women will be randomly assigned to one of two experimental conditions (n=75 per condition): 1) receiving a 10,000 steps/day recommendation and 3 health education sessions or 2) receiving an adaptive recommendation and an obesity prevention intervention. The adaptive step recommendation will update participants' recommended step counts, starting at 7,000 steps/day, then 8,000 steps/day, then finally 10,000 steps/day. Participants in the adaptive recommendation group will be provided with 3 educational sessions and will be asked to report their daily progress on weight maintenance goals via text message.

Participants will be provided pedometers and will be asked to wear them every day of the 24-week trial period.

Assessments (including self-report survey and anthropometric measurements) will be conducted at baseline, 12 weeks and 24 weeks post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 25 and over
* BMI 25 and over
* English fluency
* Not currently pregnant
* No restrictions to ambulatory activity

Exclusion Criteria:

* Current pregnancy
* Childbearing in the past 12 months
* History of myocardial infarction or stroke in last 2 years

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adherence to the pedometer-based physical activity regimen | 24 weeks post baseline

SECONDARY OUTCOMES:
Change in physical activity | 24 weeks post baseline
Change in BMI | 24 weeks post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gary Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Result] Steinberg DM, Levine EL, Askew S, Foley P, Bennett GG. Daily text messaging for weight control among racial and ethnic minority women: randomized controlled pilot study. J Med Internet Res. 2013 Nov 18;15(11):e244. doi: 10.2196/jmir.2844. PMID 24246427